CLINICAL TRIAL: NCT03052959
Title: Building on Existing Tools To Improve Chronic Disease Prevention and Screening in Public Health: Durham
Brief Title: BETTER HEALTH: Durham
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Durham Region Health Department (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-231
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cancer and Chronic Disease Prevention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental)
  Interventions: Behavioral: Immediate Intervention
- Wait List Intervention (Other)
  Interventions: Other: Wait List Intervention

INTERVENTIONS:
Behavioral: Immediate Intervention — The 'BETTER' prevention practitioner intervention involves assessment of a person's current participation, or lack of participation, among domains of evidence-based chronic disease prevention and surveillance (CDPS) actions. The assessment is followed several days later by a supportive meeting with a prevention practitioner nurse, using principles of shared decision making and health coaching, to establish goals for accomplishing CDPS activities of the individual's choice during the subsequent six months to develop personal goals and targets for participating in CDPS actions during the following six months. In BETTER HEALTH: DURHAM, the prevention practitioner nurse will be a public health nurse from the Durham Region Health Department.
  Arms: Immediate Intervention
Other: Wait List Intervention — The control arm will receive the prevention practitioner intervention 6 months after the intervention arm. Their outcomes will not be assessed in the study.
  Arms: Wait List Intervention

SUMMARY:
The BETTER intervention consists of supportive meetings between a specially trained prevention practitioner nurse and individuals aged 40-64 years to review recommended chronic disease prevention and screening activities (CDPS). The prevention practitioner nurse will assist participants to identify goals for accomplishing CDPS activities in the next 6 months. Promotion, recruitment of participants and delivery of the BETTER intervention will be adapted to meet the needs of the residents through the use of participatory research methods and community engagement strategies. The study population consists of individuals aged 40-64 years living in 10 designated areas or "clusters" within Durham Region in Oshawa and Whitby.

Objectives:

1. Help people in the designated areas identify personal goals related to chronic disease prevention and screening activities.
2. Evaluate whether the prevention practitioner was effective in helping people achieve their goals and explore whether this type of intervention could work in other settings.
3. Share what the investigators learn with government and other public health units in Ontario and across Canada.

Some clusters will receive the BETTER intervention right away and other clusters will be in a wait-list control group to receive the intervention 6 months later. Our main outcome is the change in a score that considers the number of preventive health items a person has achieved during the 6 months. The investigators will also be doing in-depth interviews and focus groups with health care providers, community organizations and people who live in the designated areas to understand whether the primary practitioner was effective.

DETAILED DESCRIPTION:
Research has shown that many Ontarians do not participate in all the chronic disease prevention and screening activities that could keep them healthy. Previous studies have found that a prevention practitioner, a nurse who works with health care providers and their practices, can be effective at improving the uptake of chronic disease prevention and screening activities.

The goal of this study is to adapt the BETTER intervention from a health care setting with family practice teams to a community-based strategy in designated areas in Durham Region. The BETTER intervention consists of supportive meetings between a specially trained prevention practitioner nurse and individuals aged 40-64 years to review recommended chronic disease prevention and screening activities (CDPS). The prevention practitioner nurse will assist participants to identify goals for accomplishing CDPS activities in the next 6 months. Promotion, recruitment of participants and delivery of the BETTER intervention will be adapted to meet the needs of the residents through the use of participatory research methods and community engagement strategies.

Previous work by the researchers identified census dissemination areas in Ontario with: (1) the lowest quintile of median household income, (2) low cancer screening rates, and 3) poor access to primary care services. The study population consists of individuals aged 40-64 years living in 10 designated areas or "clusters" within Durham Region in Oshawa and Whitby. The investigators will be working closely with local community agencies and primary care providers to identify people who may benefit from this study.

Objectives:

1. Help people in the designated areas identify personal goals related to chronic disease prevention and screening activities.
2. Evaluate whether the prevention practitioner was effective in helping people achieve their goals and explore whether this type of intervention could work in other settings.
3. Share what the investigators learn with government and other public health units in Ontario and across Canada.

Some clusters will receive the BETTER intervention right away and other clusters will be in a wait-list control group to receive the intervention 6 months later. The investigators will compare the two groups. The study will involve about 120 residents in 10 designated areas. Our main outcome is the change in a score that considers the number of preventive health items a person has achieved during the 6 months. The investigators will also be doing in-depth interviews and focus groups with health care providers, community organizations and people who live in the designated areas to understand whether the primary practitioner was effective.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40 - 64 years living in sampled low income clusters in Durham region who are English speakers (including illiterate persons). Only one participant per residential household may participate.

Exclusion Criteria:

* Unable to provide informed consent

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Paszat, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Durham Region Health Department, Whitby, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Brien MA, Lofters A, Wall B, Elliott R, Makuwaza T, Pietrusiak MA, Grunfeld E, Riordan B, Snider C, Pinto AD, Manca D, Sopcak N, Cornacchi SD, Huizinga J, Sivayoganathan K, Donnelly PD, Selby P, Kyle R, Rabeneck L, Baxter NN, Tinmouth J, Paszat L. Adaptation and qualitative evaluation of the BETTER intervention for chronic disease prevention and screening by public health nurses in low income neighbourhoods: views of community residents. BMC Health Serv Res. 2024 Apr 4;24(1):427. doi: 10.1186/s12913-024-10853-z. PMID 38575938
- [Derived] Lofters AK, O'Brien MA, Sutradhar R, Pinto AD, Baxter NN, Donnelly P, Elliott R, Glazier RH, Huizinga J, Kyle R, Manca D, Pietrusiak MA, Rabeneck L, Riordan B, Selby P, Sivayoganathan K, Snider C, Sopcak N, Thorpe K, Tinmouth J, Wall B, Zuo F, Grunfeld E, Paszat L. Building on existing tools to improve chronic disease prevention and screening in public health: a cluster randomized trial. BMC Public Health. 2021 Aug 3;21(1):1496. doi: 10.1186/s12889-021-11452-x. PMID 34344340
- [Derived] Paszat L, Sutradhar R, O'Brien MA, Lofters A, Pinto A, Selby P, Baxter N, Donnelly PD, Elliott R, Glazier RH, Kyle R, Manca D, Pietrusiak MA, Rabeneck L, Sopcak N, Tinmouth J, Wall B, Grunfeld E. BETTER HEALTH: Durham -- protocol for a cluster randomized trial of BETTER in community and public health settings. BMC Public Health. 2017 Sep 29;17(1):754. doi: 10.1186/s12889-017-4797-3. PMID 28962558

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Neighbourhoods
Period: Overall Study
Arm/Group | Immediate Intervention | Wait List Intervention
Started | 59; 5 Neighbourhoods | 66; 5 Neighbourhoods
Completed | 55; 5 Neighbourhoods | 61; 5 Neighbourhoods
Not Completed | 4; 0 Neighbourhoods | 5; 0 Neighbourhoods
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Wait List Intervention: Wait List Intervention: The control arm will receive the prevention practitioner intervention 6 months after the intervention arm.
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Wait List Intervention | Total
Number analyzed (Participants) | 59 | 66 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (6.4) | 53.2 (6.6) | 53.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 32 | 53
  Male | 38 | 34 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White | 50 | 52 | 102
  Race/ethnicity: Other | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome Measure: Mean Percentage of CDPS Actions at Baseline That Are Subsequently Met at Follow-up
Description: The primary outcome measure is the mean percentage of the number of eligible CDPS actions at baseline that are subsequently met (by self-report) at follow-up, measured at the patient level. As a function of baseline characteristics, certain individuals are eligible for certain CDPS actions. At follow-up, each patient will be re-evaluated and the number of eligible actions met will be enumerated. Six months after the baseline survey interview, the research assistant will administer the outcome survey on health and CDPS actions to participants in intervention and control clusters alike. All outcomes are self-reports of the completion of CDPS actions.
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: percent of actions
Arm/Group | Immediate Intervention | Wait List Intervention
Number analyzed (Participants) | 59 | 66
percent of actions | 64.5 (27.5) | 42.1 (23.8)

2. Secondary Outcome: Completion of Individual Actions
Description: The investigators will report the frequency with which individual CDPS actions were completed, for those actions for which the individual was eligible at baseline
Time Frame: Six months
Measure: Number; unit: percentage of eligible actions
Arm/Group | Immediate Intervention | Wait List Intervention
Number analyzed (Participants) | 59 | 66
percentage of eligible actions
  Fasting blood sugar/A1C screen | 29.0 | 25.0
  Blood pressure screen | 81.8 | 41.7
  Blood pressure monitor | 66.7 | 66.7
  LDL measured | 31.6 | 26.3
  Breast screening | 50 | 0
  Colorectal screening | 14.3 | 0
  Cervical screening | 25 | 11.1
  Body mass index screening | 72.7 | 0
  Waist circumference | 73.6 | 1.6
  Weight control | 53.8 | 57.1
  Referral for body mass index greater than 25 | 76.9 | 46.9
  Smoking cessation | 11.1 | 3.6
  Smoking cessation referral | 59.3 | 32.1
  Alcohol control | 66.7 | 52.4
  Alcohol cessation referral | 40 | 9.5
  Physical activity improved | 62.2 | 64.3
  Physical activity referral | 71.1 | 41.1
  Healthy diet score improved | 90.4 | 91.8
  Nutrition referral | 67.3 | 29.5

3. Secondary Outcome: Number of Self-referrals
Description: The investigators will report the frequency with which self-referrals were reported to the prevention practitioner.
Time Frame: Six months
Measure: Number; unit: percentage of eligible actions
Arm/Group | Immediate Intervention | Wait List Intervention
Number analyzed (Participants) | 59 | 66
percentage of eligible actions
  Fasting blood sugar/A1C screen | 29.0 | 25.0
  Blood pressure screen | 81.8 | 41.7
  Blood pressure monitored | 66.7 | 66.7
  LDL measured | 31.6 | 26.3
  Breast cancer screening | 50 | 0
  Colorectal cancer screening | 14.3 | 0
  Cervical screening | 25.0 | 11.1
  Weight control | 53.8 | 57.1
  Referral for body mass index greater than 25 | 76.9 | 46.9
  Smoking cessation referral | 59.3 | 32.1
  Alcohol cessation referral | 40 | 9.5
  Physical activity referral | 71.1 | 41.1
  Nutrition referral | 67.3 | 29.5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Immediate Intervention | Wait List Intervention
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/66
Other Adverse Events (participants affected / at risk) | 0/59 | 0/66

LIMITATIONS AND CAVEATS:
Research coordinator administering survey to participants may have served as a co-intervention; relied exclusively on self-report; excluded non-English speakers; did not explore the role of other sociodemographic characteristics such as race/ethnicity and immigration status that may intersect with income; did not explicitly compare the clusters based on factors that may have affected uptake of recommendations, such as proximity to primary care or access to public transportation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03052959/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03052959/SAP_001.pdf